CLINICAL TRIAL: NCT06469294
Title: Evaluation of Chlorhexidine Gel Associated with Photodynamic Therapy in the Treatment of Chronic Periodontitis in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, Gabriela Alessandra da Cruz Galhardo Camargo, Universidade Federal Fluminense
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 68360623.6.0000.5626; 6.019.190 (Registry Identifier: Gabriela Alessandra da Cruz Galhardo Camargo)
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Periodontitis, Adult; Periodontitis
Keywords: laser therapy; photodynamic therapy; chlorhexidine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Periodontitis; Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Clinical, laboratory, longitudinal split-mouth study carried out in humans.
Who Masked: Participant, Investigator
Masking Description: the material that will be deposited, in this case, gels for the control and placebo groups will be masked by aluminum foil for research. Gels will be encoded in a syringe and applied by researcher blind to the sites and reagents, each 4 sites will receive one og the following treatments: 1 -photodynamic therapy with red laser and photosesitization with 0,005% AM gel + 2% chlorhexidine (Fórmula e Ação Farmácia, São Paulo, SP, Brazil), 2: gel saline + lasertherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (T) - Photodynamic therapy and 2% chlorexidine and 0,005% methylene blue (Experimental): After conventional periodontal treatment, photosensitization will be performed with 2% chlorhexidine gel with 0.005% methylene blue (Fórmula e Ação Farmácia, São Paulo, SP, Brasil) for 5 minutes and photodynamic therapy will be applied with a rede laser (660nm) usinf DuoⓇ laser (MMOptics, São Carlos, SP, Brazil) with the optical fiber inside the periodontal pocket in back and forth movements, according to the manufacturer's protocol, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW.
  Interventions: Procedure: Control (C) - Saline Gel; Procedure: Test (t) - Photodynamic therapy and 2% chlorexidine and 0,005% methylene blue
- Control (C) - Saline Gel (Placebo Comparator): After conventional periodontal treatment, saline gel will be applied in the periodontal pocket and, after 5 minutes, the laser application will be simulated with the device in inactive mode, in order to maintain blinding of the patients. Application of the gel for 5 minutes and photodynamic therapy will be applied with a rede laser (660nm) usinf DuoⓇ laser (MMOptics, São Carlos, SP, Brazil) with the optical fiber inside the periodontal pocket in back and forth movements, according to the manufacturer's protocol, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW
  Interventions: Procedure: Control (C) - Saline Gel; Procedure: Test (t) - Photodynamic therapy and 2% chlorexidine and 0,005% methylene blue

INTERVENTIONS:
Procedure: Control (C) - Saline Gel — After conventional periodontal treatment, saline gel will be applied in the periodontal pocket and, after 5 minutes, the laser application will be simulated with the device in inactive mode, in order to maintain blinding of the patients.
Procedure: Test (t) - Photodynamic therapy and 2% chlorexidine and 0,005% methylene blue — After conventional periodontal treatment, photosensitization will be performed with 2% chlorhexidine gel with 0.005% methylene blue (Fórmula e Ação Farmácia, São Paulo, SP, Brasil) for 5 minutes and photodynamic therapy will be applied with a rede laser (660nm) usinf DuoⓇ laser (MMOptics, São Carlos, SP, Brazil) with the optical fiber inside the periodontal pocket in back and forth movements, according to the manufacturer's protocol, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW.

SUMMARY:
The objective of this clinical trial is to evaluate chlorhexidine gel associated with photodynamic therapy in the treatment of chronic periodontitis in Type 2 diabetics

The main questions it aims to answer are:

• To evaluate if the use of 2% chlorhexidine gel associated with 0.005% methylene blue and laser therapy is superior to conventional periodontal treatment associated with photodynamic therapy in Type 2 diabetics

Participants will receive periodontal treatment carried out with the use of 2% chlorhexidine gel associated with 0.005% methylene blue and laser therapy, associated with conventional periodontal treatment, as well as the use of photodynamic therapy associated to conventional periodontal treatment in Type 2 diabetics patientes. So, 20 periodontitis patients will be selected. Patients will be separated in two groups; Test, use of 2% chlorhexidine gel associated with 0.005% methylene blue and laser therapy + Periodontal Disease with PD> 5mm and Control, conventional periodontal treatment with gel control with fisiological solution + Laser therapy. Clinical parameters and microbiological parameters were evaluated at baseline and 3 months after periodontal treatment: Plaque Index, Bleeding On Probe, Probing depth, Gingival Recession and Clinical Attachment Level, and Microbiological parameters will be checked by PCR, for evaluating A.a, P.g., T.f., C.albicans.

DETAILED DESCRIPTION:
Periodontal disease is a polymicrobial inflammatory condition caused by infection of periodontal tissues resulting from the accumulation of bacterial biofilm, which can result in the progressive loss of the conjunctival attachment and alveolar bone. The destructive nature of diseases and their progression depend on the composition of the supra and subgingival biofilm. In response to the imbalance between host and microorganisms, the host can respond to biofilm products by generating periodontal infection. This process can result in the production of enzymes and other endogenous mediators of the inflammatory response, being responsible for much of the tissue destruction observed through clinical and histopathological parameters.

Non-surgical periodontal therapy, performed using the conventional method, tooth scaling and root planing, represents a prerequisite for the control of periodontal infections and, in most cases, is sufficient to restore periodontal health. However, some factors may be present and associated with the failure of mechanical therapy, which may be related to failure to eliminate pathogens, due to difficulty in accessing the scalers to the base of the periodontal pocket, root anatomical variations, or systemic factors that modify the response. of the host.

An important risk factor for periodontal disease is diabetes. It affects oral health and may be one of the causes for the increase in cases of tooth loss. The risk of diabetic participants having periodontitis is approximately three times greater than that of healthy participants. Diabetes can trigger an increase in the inflammatory response to the oral microbiota and can impair the host's immune response, thereby creating advanced conditions for the development and worsening of periodontal diseases in predisposed participants. At the same time, periodontitis is responsible for increasing insulin resistance and can increase the risk of diabetes or promote an impairment of glucose tolerance mechanisms. Given the bidirectional transparency between diabetes and periodontitis, it has been demonstrated that non-surgical periodontal treatment (NSPT) in participants with periodontitis and diabetes can influence glycemic control.

For the treatment of periodontal disease, surgical or non-surgical periodontal therapy is used as a basis, which aims to reduce the infection caused by dental plaque. But laser therapy is currently used as an adjuvant treatment in cases of periodontitis. The use of low-power lasers and photosensitizers has improved the reduction of bone loss and elimination of pathogenic bacteria, in addition to decontaminating periodontal pockets with almost no damage.

The direct benefits of the study are the treatment and resolution of periodontal disease for the participant and for the scientific community to indicate new forms of periodontal therapy using these medications associated with periodontal instrumentation. All tooth pocket sites in all groups will receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old
* Adults with type 2 diabetics
* Adults with periodontal disease
* Pockets with probing depth greater than 5 mm.

Exclusion Criteria:

* Participants with hypersensitivity to the components of chlorhexidine gel or methylene blue and laser therapy
* Drugs ( alcoholics, anti-inflammatories and antibiotics in the last 6 months)

Any evidence of systemic modifying factors of periodontal disease, except diabetics, and which, therefore, may directly interfere with the completion of the work. The factors described in the literature include:

* osteoporosis types I and II
* acquired or induced immunosuppression
* Pregnant or lactating women
* clinical manifestations of oral candidosis
* anti-inflammatories or hormone replacement therapy
* physical/emotional stress, medications that influence periodontal tissues.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
glycemic control | Baseline and 3 months after
  Glycemic control is the optimal serum glucose concentration in diabetic patients. It is necessary to identify factors affecting the glycemic control of patients to prevent control and complications.
  The American Diabetes Association (ADA) recommends that a HbA1c level of less than 7.0% indicates glycemic control for most adults with diabetes.
Plaque index (IP) | Baseline and 3 months after
  Plaque index are used to evaluate the level and rate of plaque formation on tooth surfaces
Clinical Attachment Level (CAL) | Baseline and 3 months after
  CAL represents the extent of periodontal support that has been lost around a tooth and is measured with the periodontal probe as the distance from the cemento-enamel junction (CEJ) to the base of the pockesites per tooth, from cementoenamel junction to gingival margin, using periodontal probe < 3mm indicate good results.
Pocket Probing Depht (PPD) | baseline and 3 months after
  Probing depth (referred to as pocket depth if periodontal disease is present) is the distance from the gingival margin to the apical portion of the gingival sulcussites per tooth using a periodontal probe. The PPD corresponds to the distance from the gingival margin to the apical portion of the gingival sulcus or periodontal pocket. Less than or equal to 3 millimeters
Bleending on Probing (BOP) | baseline and 3 months ago
  Bleeding on probing (BOP) is the primary parameter to set the threshold for gingivitis and is recorded using the gingival index score (GI). Less than 10% of bleeding sites.
Clinical Recession | Baseline and 3 months after
  Gingival recession is the exposure of the root surface resulting from migration of the gingival margin apical to the cementoenamel junction (CEJ).
glycated hemoglobin | Baseline and 3 months after
  Glycated hemoglobin, also known as HbA1c, glycohemoglobin, glycosylated hemoglobin, or simply A1c. HbA1c is measured primarily to determine the three-month average blood sugar level and can be used as a diagnostic test for diabetes mellitus and as an assessment of glycemic control. The American Diabetes Association (ADA) recommends an HbA1c level of less than 7.0% as a glycemic target for nonpregnant adults with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela AC Camargo, doctor, Principal Investigator — University Federal Fluminense
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
The result will be communicated verbally to each participant.

REFERENCES:
- [Background] Corbella S, Calciolari E, Donos N, Alberti A, Ercal P, Francetti L. Laser treatments as an adjunct to non-surgical periodontal therapy in subjects with periodontitis and type 2 diabetes mellitus: a systematic review and meta-analysis. Clin Oral Investig. 2023 Apr;27(4):1311-1327. doi: 10.1007/s00784-023-04873-y. Epub 2023 Feb 28. PMID 36849595